CLINICAL TRIAL: NCT05872464
Title: Efficacy and Safety of Artificial Saliva Containing Cumin and Ginger Extract in Head and Neck Cancer Patients With Xerostomia
Brief Title: Artificial Saliva Containing Cumin and Ginger Extract in Head and Neck Cancer Patients With Xerostomia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chulalongkorn University (Other)
Responsible Party: Principal Investigator, Pornanong Aramwit, Pharm.D., Ph.D, Professor, Chulalongkorn University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R177h/66
Record Dates: First submitted 2023-05-11; First posted 2023-05-24 (Actual); Last update posted 2024-06-24 (Actual); Status verified 2024-06

CONDITIONS: Xerostomia
MeSH Terms: conditions — Xerostomia | interventions — ginger extract

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Artificial saliva containing cumin and ginger extract (Experimental): Artificial saliva containing cumin and ginger extract in spray bottle
  Interventions: Other: Artificial saliva containing cumin and ginger extract
- Placebo (Placebo Comparator): Placebo containing composition close to the test group without cumin and ginger extract in spray bottle
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Artificial saliva containing cumin and ginger extract — Artificial saliva containing cumin and ginger extract in spray bottle
  Arms: Artificial saliva containing cumin and ginger extract
Other: Placebo — Placebo containing composition close to the test group without cumin and ginger extract in spray bottle
  Arms: Placebo

SUMMARY:
The objectives of this study are to evaluate efficacy and safety of artificial saliva containing cumin and ginger extract in head and neck cancer patients with xerostomia.

DETAILED DESCRIPTION:
There are 52 patients in this study. They are divided into 2 groups which are artificial saliva containing cumin and ginger extract group (test group) 26 patients and placebo group 26 patients. The patients spray the sample into the mouth 3 times/day for 14 day. Amount of saliva, pH of saliva, xerostomia questionnaires, WHO Oral Mucositis Grading Scale, quality of life, adverse events, and satisfaction were assessed.

ELIGIBILITY:
Inclusion Criteria:

* Age more than 18 years
* Head and neck cancer with xerostomia
* 6 months post radiation
* Willing to participate in this study

Exclusion Criteria:

* Sialolith or Sjogren's syndrome
* Uncontrolled cancer
* Using artificial saliva more than 2 weeks
* Taking Pilocarpine or cevimeline more than 2 weeks
* Allergic to cumin, ginger, xylitol, and glycerin
* History of other oral mucosal diseases
* Pregnancy and lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2025-05-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Amount of saliva | 14 days
  Spit saliva to the bottle for 5 min

SECONDARY OUTCOMES:
Acid and base characteristic of saliva | 14 days
  Spit saliva to the bottle, then take 1 piece of pH strip and dip it into the saliva for 30 seconds. Compare the color of the dipped pH strip to the color chart on pH strip box. The result shows value at pH 1-14.
Xerostomia questionnaires | 14 days
  Assessment xerostomia symptom by patient (scoring 1 to 10 point (low to high xerostomia severity)).
Oral Mucositis Grading Scale | 14 days
  Evaluate oral mucosa by physician (scoring 0 to 4 point (none to life-threatening)).
Adverse reaction: Skin reaction | 14 days
  Found or not found
Adverse reaction: Respiratory reaction | 14 days
  Found or not found
Adverse reaction: Gastrointestinal trat reaction | 14 days
  Found or not found
Quality of life of the patient | 14 days
  Assessment quality of life by patient (scoring 1 to 120 point (high to low quality of life)).
Satisfaction of the patient | 14 days
  Assessment satisfaction by patient (scoring 1 to 10 point (low to high satisfaction)).

CONTACTS AND LOCATIONS:
Overall Officials: Pornanong Aramwit, Professor, Principal Investigator — Chulalongkorn University